CLINICAL TRIAL: NCT04804501
Title: Effect of Blue Light Glasses on Screen Usage After a Concussion in College Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rochester Institute of Technology (Other)
Responsible Party: Principal Investigator, Zachary Bevilacqua, Principal Investigator, Rochester Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RochesterIT
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Brain Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Blue Light Glasses (experimental) (Experimental): These subjects will wear the device (glasses) while performing a reading task.
  Interventions: Device: Blue Light Glasses; Other: Computer Reading Task
- No Glasses (control) (Other): These subjects will not wear the device (glasses) while performing a reading task.
  Interventions: Other: Computer Reading Task

INTERVENTIONS:
Device: Blue Light Glasses — Participants will be randomized into an experimental group (blue light glasses) or a control group (no glasses). Participants will perform a computer reading task while either wearing, or not wearing the glasses.
  Arms: Blue Light Glasses (experimental)
Other: Computer Reading Task — Participants will read on a computer until concussion symptoms increase by a score of 3 or more (reading task termination criteria). One or more points will be assigned for each increase in symptom severity, and one point will be assigned for each new symptom that appears.

SUMMARY:
Premature cessation of screen usage is a common behavior post-concussion, given the taxing nature of a screen-time task. In the academic setting, screen-time is a near unavoidable component, however, complete avoidance of class and screen use may in fact provoke psychological symptoms of anxiety and depression in students, for fear of falling behind in their studies. Thus, compensatory measures should be investigated to assist students as they attempt to maintain academic involvement throughout their concussion recovery. Blue light blocking glasses have been shown to significantly increase screen-time usage in individuals with post-concussion syndrome, yet these results are only representative of a small portion of the concussion population. Thus, we propose investigating whether blue light blocking glasses can prolong screen usage prior to symptom exacerbation, specifically in concussed students that are still within the normal recovery timeframe. This cross-sectional randomized clinical trial will provide further evidence of the utility blue light blocking glasses can offer as a therapeutic tool for students recovering from concussion. We would like to test volunteers from the Rochester Institute of Technology who have been treated by a medical provider within the university's health center. Blue light glasses will be worn during a one-time computer reading task while the subject is participating in the study. The total time for the complete the reading task is dependent upon the participant's symptom fluctuations; however, we suspect completion criteria will be met within 20 minutes from beginning. The risks in this study are minimal and results may increase our understanding of therapeutic tools for patients with ocular-driven concussion symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Full-time student at RIT
* Diagnosed mild traumatic brain injury
* Between 18-26 years of age
* Within 3-14 days post-injury

Exclusion Criteria:

* Any head, neck, or face injury in the 1 year prior to the study (e.g., concussion, eye injury) other than the current injury
* History of vestibular or ocular dysfunction\
* Any neurological disorders (e.g., seizure disorders, closed head injuries with loss of consciousness greater than 15 minutes, CNS neoplasm, history of stroke)
* Injury more severe than mild traumatic brain injury (skull fracture, positive CT or MRI)
* Having taken pain medication within 8 hours prior to testing
* Not able to personally consent
* Pregnant
* Deaf or hard of hearing.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Time on Screen | 30 minutes or less
  The amount of time a participant can spend on time, prior to meeting termination criteria, will be recorded and compared between experimental and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Rochester Institute of Technology, Rochester, New York, United States